CLINICAL TRIAL: NCT01761578
Title: First in Man Safety Evaluation of the ART18Z Bioresorbable Stent for the Treatment of Single de Novo Lesion of a Native Coronary Artery.
Brief Title: ARTDIVA Study : First in Man Safety Evaluation of the ART18Z Bioresorbable Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arterial Remodeling Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTDIVA
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
Keywords: Bioresorbable; Coronary; Stent; Vascular Remodeling; Angioplasty; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Vascular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ART18Z Bioresorbable stent (Experimental)
  Interventions: Device: ART18Z Bioresorbable stent

INTERVENTIONS:
Device: ART18Z Bioresorbable stent — The drug free fully bioresorbable coronary stent ART18Z is a balloon expandable poly lactic acid stent.

SUMMARY:
This prospective, multicentre, open labeled, single arm, first in man interventional investigation aims to evaluate the safety of the ART18Z bioresorbable stent for the treatment of patients with single de novo lesion of a native coronary artery with mandatory balloon predilatation.

ELIGIBILITY:
Eligibility:

- Healthy voluntary and women of child-bearing potential are not accepted

Inclusion Criteria:

Angiographic Inclusion Criteria:

Target lesion must meet all of the following criteria

* Single vessel lesion
* De novo lesion
* Located in a native coronary artery with visually estimated nominal artery diameter of 2.8 to 3.2 mm
* Length ≤ 8 mm visually estimated
* Located in a major artery or branch with a visually estimated stenosis >50% and <100% with a TIMI flow ≥1

General Inclusion Criteria:

Patient profile:

* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the ART18Z Bioresorbable Stent.
* Patient provides written informed consent approved by the EC prior to any clinical investigation related procedure
* Patient must agree to undergo all clinical investigation plan - required clinical follow-up visits, QCA, OCT
* Patient must agree not to participate in any other clinical investigation for a period of 3 years following the procedure
* a social security number is required, otherwise patients cannot be included in the trial.

Clinical profile:

* Silent ischemia, stable or unstable angina with documented ischemia (stress echocardiography, 12-lead ECG, nuclear imaging, bicycle test, Treadmill stress test)
* 3 months limited clopidogrel treatment must be acceptable in compliance with patient health status
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery

Exclusion Criteria:

Angiographic Exclusion Criteria:

* Target lesion meets any of the following criteria:
* Aorto-ostial location (within 3 mm)
* Left main location
* located within 3 mm of the origin of the LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and >20% stenosed lesion, by visual estimation) arterial or saphenous vein graft
* Lesion involving a bifurcation ≥ 1.5 mm in diameter and ostial lesion > 40% stenosed by visual estimation or side branch requiring predilatation
* Excessive tortuosity proximal to or within the lesion (Extreme angulation (≥ 90%) proximal)
* Calcification lesion
* Restenotic from previous intervention
* The target vessel contains visible thrombus
* Chronic total occlusion (CTO)
* Another clinically significant lesion is located in the same major epicardial vessel as the target lesion (including side branches)
* Patient has a high probability that a procedure other than pre-dilatation and stenting will be required at the time of procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon)
* Non clinical investigation percutaneous intervention in the target vessel < 6 months prior to or if planned to be done within 6 months after the investigational procedure.
* Non clinical investigation percutaneous intervention in a non-target vessel < 1 months prior to the investigational procedure with TIMI flow = 3 and no evidence of dissection at the time of the clinical investigation procedure, or if planned to be done within 6 months after the investigational procedure.

General Exclusion Criteria

* Evidence of an acute MI within 3 weeks of the intended investigational procedure
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction (LVEF) < 30%
* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
* Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Patient has known renal insufficiency with creatine clearance < 40 ml/min or patient on dialysis
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebro vascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a < 24 months limited life expectancy
* Vulnerable population (refer to §6.4)
* Patient is already participating in another clinical investigation that has not yet reached its primary endpoint
* Pregnant or nursing patients and those who plan pregnancy during the clinical investigation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
MACE rate | at 6 months
  Major Adverse Cardiac Event is defined as death, MI (Myocardial Infarction) or any TLR (Target Lesion Revascularization).

SECONDARY OUTCOMES:
Acute Performances (Device/Procedure Success) | Procedure and post-procedure up to 24 hours
Stent thrombosis | at 1, 3, 6, 12, 18 months
Clinically driven TVF, TLR, TVR | at 1, 3, 6, 12, 18 months
Evolution of Angiographic binary restenosis | at 12 months
Evolution of Angiographic in-stent Late Lumen Loss | at 12 months
Percentage of stent coverage by OCT | at 12 months
Evolution of the neointima by OCT | at 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Polyclinique les Fleurs, Ollioules
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Haut Leveque, Pessac
  - Clinique Pasteur, Toulouse
  - Hôpital Rangueil, Toulouse

REFERENCES:
- See also: Related Info — http://www.art-stent.com